CLINICAL TRIAL: NCT03754062
Title: Pharmacological Modulation of Belief Salience
Acronym: MOBS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HR-16/17-0603
Record Dates: First submitted 2018-10-23; First posted 2018-11-27 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-02

CONDITIONS: Haloperidol; Placebo; L-DOPA
MeSH Terms: interventions — Levodopa; Haloperidol

STUDY DESIGN:
Intervention Model Description: Placebo x Haloperidol x LDOPA
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo - Cap
- Haloperidol 3mg (Experimental): Haloperidol
  Interventions: Drug: Haloperidol
- L-Dopa 150 mg & Domperidone 10mg (Experimental): L-Dopa
  Interventions: Drug: L-dopa

INTERVENTIONS:
Drug: Placebo - Cap — Administration of Placebo by pill.
  Arms: Placebo
Drug: L-dopa — Administration of L-dopa by pill.
  Arms: L-Dopa 150 mg & Domperidone 10mg
Drug: Haloperidol — Administration of Haloperidol by pill.
  Arms: Haloperidol 3mg

SUMMARY:
To provide an initial test of the hypothesis that dopamine mediates the motivational salience of stimuli beyond simple stimulus-reinforcement associations, the researchers propose to undertake a study of the modulation of a) levels of agreement or disagreement with; b) the perceived self- relevance; and c) the perceived interest of propositions expressing beliefs and values in healthy male volunteers using Ii) a dopamine antagonist (the D2-blocker haloperidol), and (ii) a dopamine precursor L-Dopa to increase CNS dopamine transmission.

The researchers will also administer the Salience Attribution Task (SAT) which will allow researchers to assess reward-learning processing of simple stimuli using a reaction-time game. This task was utilised by Roiser et al in order to explore whether delusions in medicated patients with schizophrenia were related to impairments in associative learning. The authors hypothesised that associative learning was influenced by D2 receptor blockade. The researchers extend this approach to examine the effect of dopamine modulation on the SAT as a measure of associative learning, a basic neuropsychological process that may be involved in the attribution of salience to beliefs.

Finally, the researchers will ask participants to perform a within-subjects dictator game to understand the influence of dopaminergic manipulation of the live attribution of harm intention to partners. The task has been previously validated online. Participants will play against 3 partners in a random order in each drug condition. Each partner will play the participant for 6 trials. One partner will always be fair, one will always be unfair, and one will be 50% unfair. We aim to understand whether potentiating dopamine has an additive effect on the harm intention attributions toward partners, regardless of the behaviour of the partner.

DETAILED DESCRIPTION:
Delusions in psychiatry are viewed as a form of aberrant belief. Consequently it is important to understand the cognitive and neural processes involved in beliefs to provide insights into how these processes go awry in the formation of delusions. Beliefs have been defined as 'a disposition to express, assent to, or otherwise act in accordance with some proposition'. Some beliefs are widely held within a given society (e.g the earth revolves around the sun; eating humans is wrong), whereas others vary in association with subcultural and individual differences (e.g God created the universe; abortion is wrong). Similarly, the conviction or agreement with which an individual's beliefs and values are held may change over time, to the extent that some beliefs and values may be lost, and others acquired. Also, the perceived relevance of beliefs and values to oneself may vary. For example, beliefs that the 'earth revolves around the sun' and that 'global warming is occurring' may both be held with conviction, but the latter may be perceived as having higher relevance to the self in terms of risk, and potential life-style changes. Hence, self-relevance is a dimension of beliefs that is potentially dissociable from the conviction (level of agreement) with which a belief is held. Further, some propositions expressing beliefs and values may be regarded as more interesting than others. This raises the question of what neurobiological processes contribute to the sense of conviction for, and perceived self-relevance and interest of beliefs and values?

The mesolimbic dopamine system is a candidate neural system implicated in mediating the motivational salience of perceptions and ideas, 'whereby events and thoughts come to grab attention, drive action, and influence goal-directed behaviour because of their association with reward or punishment'. In human studies, haloperidol has been used to show that dopamine activity influences action-value estimates represented in the striatum during instrumental conditioning, as would be expected from earlier studies of feedback-based learning. Still other data suggest that brain regions rich in dopaminergic inputs play a role in processing the salience of rewarding events. What is not known is if these dopaminergic rich regions also modulate the motivational salience of more complex 'stimuli' including ideas and beliefs.

Main hypothesis:

Prediction 1:

At a neurobiological level, the hypothesis is that the mesolimbic dopamine system is recruited to tag representations (ideas and beliefs) as motivationally salient. Potentiation of dopamine transmission should increase salience of beliefs (as indicated by increases in agreement, self-relevance and interest toward propositions within science, paranormal, politics, moral, and religious themes in the Beliefs and Values Inventory while attenuation of dopamine transmission should be associated with decreased salience. Answers of items within themes will be summed to create summary scores that will be split by agreement, interest, and self-relevance dimensions.

Prediction 2:

Potentiating dopamine be associated with increased attribution of harmful intent to partners across all trials (but trait paranoia will not be associated with variation in attributions of self-interest) of a within-subjects dictator game.

Prediction 3:

Attribution of harmful intent to different dictators will follow a dose-response relationship (fair < partially fair < unfair) across all ranges of dopamine potentiation. However, L-Dopa conditions will have a higher baseline of average harmful intent. There will be no interaction between dopamine manipulations and dictator fairness on attribution of harmful intent.

If these hypotheses receive empirical support, it would be relevant to understanding the role of the dopamine system in normal cognitive processes involved in expressing or acting in accordance with beliefs. It would also be relevant to determining the role of dopamine dysregulation in psychosis (in delusion formation). Also, reduced levels of the meaningfulness of experience following antipsychotic administration (as indexed by reduced agreement for and perceived self- relevance and interest of beliefs and values) would identify a potential reason for non-compliance with antipsychotic treatment.

Supplementary hypotheses:

There will be an interaction between condition (placebo, dopamine blockade, dopamine potentiation) x dimension (agreement, self-relevance, interest), whereby self-relevance and interest are affected more by dopamine modulation than agreement. This might explain why patients with delusions who are given antipsychotics will continue to say that they believe 'x,' but don't think about it as much, and cease to act upon it.

Aims:

To provide an initial test of the hypothesis that dopamine mediates the motivational salience of stimuli beyond simple stimulus-reinforcement associations, we propose to undertake a study of the modulation of a) levels of agreement or disagreement with; b) the perceived self- relevance; and c) the perceived interest of propositions expressing beliefs and values in healthy male volunteers using i) a dopamine antagonist (the D2-blocker haloperidol), and (ii) a dopamine precursor L-Dopa to increase CNS dopamine transmission.

The researchers will also administer the Salience Attribution Task (SAT) which will allow the researchers to assess reward-learning processing of simple stimuli using a reaction-time game. This task was utilised by Roiser et al. in order to explore whether delusions in medicated patients with schizophrenia were related to impairments in associative learning. The authors hypothesised that associative learning was influenced by D2 receptor blockade. We extend this approach to examine the effect of dopamine modulation on the SAT as a measure of associative learning, a basic neuropsychological process that may be involved in the attribution of salience to beliefs.

Finally, the researchers will ask participants to perform a within-subjects dictator game to understand the influence of dopaminergic manipulation of the. Participants will play against 3 partners in a random order in each drug condition. Each partner will play the participant for 6 trials. One partner will always be fair, one will always be unfair, and one will be 50% unfair. We aim to understand whether potentiating dopamine has an additive effect on the harm intention attributions toward partners, regardless of the behaviour of the partner.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between the ages of 18-65

Exclusion Criteria:

* History or current psychiatric or neurological illness, history or current serious medical diagnosis, BMI outside of normal/healthy range, smoker over 5 cigarettes per day, recent use of drugs, non-english speaker.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Beliefs and Values Inventory (BVI) | 12 Months
  Change in score between conditions on the BVI. Scores will be summed by item totals within theme (paranormal, religion, morality, politics, and science) and dimension (agreement, self-relevance, and interest).
Salience Attribution Test (SAT) | 12 Months
  Change in attribution of explicit and implicit salience between conditions on the SAT.
Within-subjects dictator game | 12 Months
  Participants will play against three different partners, each for six trials. In each trial, the player's partner will have the option to either split or take 10p from the player, so that the player either ends up with 5p or 0p. Players will play against one partner that will always split the money, one that will always take all of the money, and one that will 50% of the time split the money. After each trial, the player will be asked on a scale of 1-100 (1 being not at all and 100 being completely):
  1. How much do you think your partner was driven by a desire to increase their own bonus, and
  2. How much do you think your partner was driven by a desire to reduce your bonus.
  Total of a. and b. will be added up for each style of partner for each arm.

SECONDARY OUTCOMES:
Big-5 Personality Questionnaire | 6 Months
  The researchers will calculate the associations between personality dimensions of the Big-5 (extraversion, neuroticism, openness, agreeableness, and conscientiousness) using the 25 item version (scores from 1-5 on a likert scale, with 5 meaning higher agreement with a statement) with variation within-subjects.
  Each dimension will be totalled to calculate personality variation.
Brief Oxford-Liverpool Inventory of Experiences and Feelings | 6 Months
  The researchers will calculate the associations between baseline schizotypy scores with variation within-subjects across conditions.
  Unusual Experiences (hallucinations etc), Cognitive Disorganisation (cognitive difficulties), Introvertive Anhedonia (loss of pleasure etc.), and Impulsive Nonconformity (impulsiveness) sub-scales will be added up individually (from a scale of 1-5 for each item, 5 being higher agreement with an item) to calculate schizotypy on a number of dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Neuroimaging Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Share anonymised data after collection on the Open Science Framework.

REFERENCES:
- [Result] Schmidt K, Roiser JP. Assessing the construct validity of aberrant salience. Front Behav Neurosci. 2009 Dec 23;3:58. doi: 10.3389/neuro.08.058.2009. eCollection 2009. PMID 20057930
- [Result] Kapur S. Psychosis as a state of aberrant salience: a framework linking biology, phenomenology, and pharmacology in schizophrenia. Am J Psychiatry. 2003 Jan;160(1):13-23. doi: 10.1176/appi.ajp.160.1.13. PMID 12505794
- [Result] Pessiglione M, Seymour B, Flandin G, Dolan RJ, Frith CD. Dopamine-dependent prediction errors underpin reward-seeking behaviour in humans. Nature. 2006 Aug 31;442(7106):1042-5. doi: 10.1038/nature05051. Epub 2006 Aug 23. PMID 16929307